CLINICAL TRIAL: NCT06264102
Title: Effect of Dalcroze Eurhythmics' Physical Exercises on Headaches, Backaches, and Leg Pains in Older Women: a Randomized Controlled Trial
Brief Title: Influence of Dalcroze Eurhythmics on Pains in Older Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024/1/1
Record Dates: First submitted 2024-01-30; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-01

CONDITIONS: Back Pain; Headache; Leg Pain
Keywords: headache; elderly women; Dalcroze Eurhythmics; back pain; leg pain
MeSH Terms: conditions — Back Pain; Headache

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Physical exercises program
  Interventions: Other: Physical exercise program
- Control group (No Intervention): Were advised not to change anything about their current lifestyle, and in particular not to undertake any new structured physical activity.

INTERVENTIONS:
Other: Physical exercise program — Training sessions took place twice a week for 45 minutes each over a period of 12 weeks. Each training included rhythmic exercises using the Jaques-Dalcroze Eurhythmics (JDE) method with piano accompaniment and electronically played music. Training sessions were conducted by a JDE specialist.
  Exercises with the use of this method consist mainly in the repetition of preset musical sequences using body movements. In addition to the physical layer, the cognitive layer was equally important: while performing a given movement exercise, participants often had to focus in order to react appropriately to additional tasks, such as changes in sound pitch and rhythm of the piece.
  Arms: Intervention group

SUMMARY:
In this study, we attempted to answer the question of whether participation in a 12-week rhythmic exercise program using the Dalcroze method affects the level of intensity of pain experienced by women over the age of 65. The level of pain was determined on a numerical scale from 1 to 10 and involved headaches, back pain and leg pain.

DETAILED DESCRIPTION:
Background. Body pain of various degrees and types can complicate human life. Regular physical exercise and good mental health can both have protective effects on the body and its physical health. Physical exercises may also, in some aspects, be particularly important for older women who experience varying degrees of headache, back pain, and/or leg pain chronically. The purpose of the study was to analyze the effects of the Dalcroze Eurhythmic Method on headaches, backaches, and leg pains among older women.

Methods. Sixty-two blinded participants with pain were randomized into two groups. Women (65 to 82 years old) who had reported the occurrence of headaches, backaches, or leg pains during the 3 months prior to the beginning of the randomized controlled trial study were identified. The participants in the pre-test and post-test used the 0-10 Numeric Pain Rating Scale to quantify their pain. Women from the experimental group participated for 3 months in the physical exercise program based on the Dalcroze Eurhythmics Method.

ELIGIBILITY:
Inclusion Criteria:

* female, 65+ years old, physical and mental state that allows them to participate in the exercise program (ability to follow the instructions), community dwelling

Exclusion Criteria:

* taking analgesics indelibly, Parkinson's or Alzheimer's disease, using social assistance or nursing care.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Pain levels before exercise program | From enrollment to the day before the start of the exercise program
  Level of pains determined by numeric pain scale 1-10

SECONDARY OUTCOMES:
Results of pain levels after exercise program | One month after completion of the exercise program
  Level of pains determined by numeric pain scale 1-10

CONTACTS AND LOCATIONS:
Overall Officials: JANUSZ MACIASZEK, PROF, Study Director — Poznan University of Physical Education
Locations (1):
- Poznan University of Physical Education, Poznan, Wielkopolska, Poland